CLINICAL TRIAL: NCT05565040
Title: Concealed Penis in Pediatric Age Group; A Comparison Between Three Surgical Techniques
Brief Title: Concealed Penis in Pediatric Age Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egyptian Biomedical Research Network (Network)
Responsible Party: Principal Investigator, Ahmed Elrouby, Associate Professor of Pediatric Surgery, Alexandria University, Egyptian Biomedical Research Network
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0305434
Record Dates: First submitted 2022-09-21; First posted 2022-10-04 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Pediatric ALL; Surgery; Urologic Diseases
Keywords: Concealed; phallopexy; dartos excision; degloving; penile re-retraction
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Urologic Diseases; Degloving Injuries | interventions — Circumcision, Male

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phallopexy group (Experimental): phallopexy only
  Interventions: Procedure: Circumcision in concealed penis
- Dartos excision group (Experimental): complete circumferential dissection and excision of dartos fascia only
  Interventions: Procedure: Circumcision in concealed penis
- Combined phallopexy and dartos excision group (Experimental): phallopexy as in patients of group A but after complete dissection and excision of dartos fascia
  Interventions: Procedure: Circumcision in concealed penis

INTERVENTIONS:
Procedure: Circumcision in concealed penis — comparison of three surgical techniques (as described in the arms) in the management of concealed penis in pediatrics

SUMMARY:
Background: Comparison between three different surgical techniques in the management of concealed penis. Methods: This prospective interventional non-randomized study included 150 pediatric patients with concealed penis. They were distributed equally into three groups; group A; patients treated by phallopexy only, group B; patients treated by complete dissection and excision of dartos fascia & group C; patients treated by both phallopexy and dartos excision.

DETAILED DESCRIPTION:
Background: Comparison between three different surgical techniques in the management of concealed penis. Methods: This prospective interventional non-randomized study included 150 pediatric patients with concealed penis. They were distributed equally into three groups; group A; patients treated by anchoring the penile skin dermis to Buck's fascia at the penile base at 3 & 9 o'clock points using PDS 5/0 (phallopexy), group B; patients treated by complete dissection and excision of dartos fascia & group C; patients treated by phallopexy as in group A after complete dissection and excision of dartos fascia. Follow-up at the end of the 1st post-operative week and then monthly for 6 months as regards penile skin congestion and/or necrosis, wound infection, edema, and/or re-retraction was carried out.

ELIGIBILITY:
Inclusion Criteria:

* patients with a buried penis at or below the pubic skin level with a stretched penile length for all of them within the normal range according to their ages as titrated in the literature

Exclusion Criteria:

* Patients with any associated anomalies like hypospadias, torsion, penoscrotal web, micropenis, mega-prepuce, or chordae were excluded from the study.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Post-operative appearance of penile skin congestion and/or necrosis | 6 months
  Repeated and regular monthly examination of the patients as regards persistent bluish penile discoloration and or loss of penile skin viability. Also a questionnaire of parents about penile skin color, loss of skin, and/or appearance of any abnormal tissues
Wound infection | 6 months
  Repeated and regular monthly examination of the patients as regards the appearance of any penile skin infection and/or pyogenic discharge. Also a questionnaire of parents about the appearance of penile skin redness, pyogenic discharge, and/or the appearance of any pyogenic membranes
Penile edema | 6 months
  Repeated and regular monthly examination of the patients as regards the appearance of penile skin edema. Also a questionnaire of parents about any increase of penile girth than the usual
Penile re-retraction | 6 months
  Repeated and regular monthly examination of the patients as regards the development of any penile re-retraction in the form of retraction of the penis to or beneath the level of pubic skin. Also, a questionnaire of parents about this finding was done

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed EZ Elrouby, A.Professor, Principal Investigator — University of Alexandria
Locations (1):
- Faulty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Elrouby A. Concealed penis in pediatric age group: a comparison between three surgical techniques. BMC Urol. 2023 Jan 11;23(1):9. doi: 10.1186/s12894-022-01169-3. PMID 36631822

DOCUMENTS (1):
  • Study Protocol (2022-01-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT05565040/Prot_000.pdf